CLINICAL TRIAL: NCT01384071
Title: The Effects of Unstable Shoes on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Armand Staphane, PhD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBP-2011
Record Dates: First submitted 2011-06-15; First posted 2011-06-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Unstable shoes; Gait; Balance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unstable shoes (MBT) (Experimental): MBT shoes (Masai Barefoot Technology, Switzerland)
  Interventions: Device: Unstable shoes (MBT)
- Stable shoes (Adidas) (Sham Comparator): Adidas stable shoes (Adidas Bigroar2)
  Interventions: Device: Sham intervention (Adidas shoes)

INTERVENTIONS:
Device: Unstable shoes (MBT) — Wearing unstable (MBT) shoes during 6 weeks
  Arms: Unstable shoes (MBT)
Device: Sham intervention (Adidas shoes) — Normal stable shoes (Adidas Bigroar2)
  Arms: Stable shoes (Adidas)

SUMMARY:
Some physicians, physiotherapists and nurses use or even suggest unstable shoes in cases of low back pain. No studies on the real effects of these shoes on low back pain in health care professions have been carried out and therefore as yet there is no real evidence of their effectiveness. Thus the investigators assume that wearing unstable shoes over a period of six weeks could reduce low back pain and functional disability due to the changes of the gait and posture and may increase the quality of life.

The purposes of this study are:

1. To evaluate the modifications of pain level, functional capacity and quality of life among individuals with moderate level of non-specific chronic low back pain after wearing unstable shoes.
2. To quantify biomechanical modifications of gait and posture.

ELIGIBILITY:
Inclusion criteria:

* employees of Geneva University Hospital
* working in a standing position for at least 50% of their working day
* aged between 30 and 65
* having chronic low back pain that has been defined at least 3 out of 10 on a visual analogue scale during the last 3 months or the need to take regular pain medication for this reason

Exclusion criteria:

* having severe pain in other body parts
* undergone back surgery, neurological or balance problems
* inability to walk a distance of 100 meters
* already worn unstable shoes and being off of work because of low back pain

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in low back pain at 6 weeks | Baseline and 6 weeks
  Low back pain level with the visual analogue scale (VAS) from 0 to 10;
Change from baseline in the Roland-Morris disability questionnaire at 6 weeks | Baseline and 6 weeks
  functional disability with the Roland-Morris disability questionnaire (this questionnaire has been validated in French as the Functional Disability Scale for the Assessment of Low Back Pain - Eifel)
Change from baseline in the EQ-5D quality of life questionnaire at 6 weeks | Baseline and 6 weeks
  Quality of life with the EQ-5D.

SECONDARY OUTCOMES:
Change from baseline in gait speed at 6 weeks | Baseline and 6 weeks
  Seft-selected gait speed
Change from baseline in balance performance at 6 weeks | Baseline and 6 weeks
  center of pressure speed in conditions :
  * eyes opened and eyes closed
  * stable and unstable surface
Change from baseline in ankle dorsiflexion during gait at 6 weeks | Baseline and 6 weeks
  Ankle dorsiflexion at initial contact during gait
Change from baseline in pelvis anteversion during gait at 6 weeks | Baseline and 6 weeks
  Mean pelvis anteversion during gait
Change from baseline in trunk anteversion during gait at 6 weeks | Baseline and 6 weeks
  Mean trunk anteversion during gait
Change from baseline in activation period of lower-limb muscles during gait at 6 weeks | Baseline and 6 weeks
  Activation period of lower-limb muscles (gasctrocnemius, peroneus, tibialis anterior, rectus femoris and semi-tendinosus) during gait
Change from baseline in activation period of erector spinae during gait at 6 weeks | Baseline and 6 weeks
  Activation period of erector spinae during gait
Change from baseline in maximum knee extension during gait stance phase at 6 weeks | Baseline and 6 weeks
  Maximum knee extension during stance phase

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland